CLINICAL TRIAL: NCT05354362
Title: An Open Label, Phase Ⅰb Study of ATG-010 in Combination With ATG-008 in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma (RR DLBCL)
Brief Title: A Study of ATG-010 in Combination With ATG-008 in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Acronym: MATCH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the adjustment of clinical research and development strategy，sponsor decided to terminate the study
Sponsor: Antengene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-008&010-DLBCL-001
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-07

CONDITIONS: Relapsed/Refractory Diffuse Large B-cell Lymphoma
Keywords: Lymphoma, Hodgkin's lymphoma , non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-010 and ATG-008 (Experimental): ATG-010 and ATG-008 should be taken 6 hours apart on a PK sampling day
  Interventions: Combination Product: ATG-010 and ATG-008

INTERVENTIONS:
Combination Product: ATG-010 and ATG-008 — Patients enrolled will receive consecutive daily treatment at assigned dose level. The starting dose of ATG-010 at the dose escalation phase will be 60 mg QW, which could be escalated to 80 mg QW, 100 mg QW, 60 mg BIW. In case 60 mg QW of ATG-010 with any dose of ATG-008 is NOT tolerable, 40 mg QW ATG-010 could be explored. The starting dose of ATG-008 will be 15 mg QD, which could be escalated to 20 mg QD, with maximum of 30 mg QD. SRC will be consulted before each dose escalation starts.

SUMMARY:
This is an Open label, Phase Ⅰb Study of ATG-010 in Combination With ATG-008 in Patients with Relapsed/Refractory Diffuse Large B-cell Lymphoma (RR DLBCL)

DETAILED DESCRIPTION:
This is a multi-center, open label, phase 1 study conducted in RR DLBCL patients. The MTD and/or RP2D of study treatment, ATG-010 in combination with ATG-008, will be selected using BOIN design for the dose escalation phase. Additional patients will be enrolled as an expansion cohort after MTD and/or RP2D is determined.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. ECOG Performance score of ≤2.
3. Estimated life expectancy of >3 months.
4. Previously treated, pathologically confirmed DLBCL
5. Patients must have received at least 2 but no more than 5 previous systemic regimens (for non-DH/TH, non-DE DLBCL and DLBCL not transformed from FL or CLL), or at least 1 but no more than 5 previous systemic regimens (for DH/TH, DE DLBCL, and DLBCL transformed from FL or CLL) for the treatment of their DLBCL.

   1. Prior stem cell transplantation is allowed; induction, consolidation, stem cell collection, preparative regimen and transplantation ± maintenance are considered a single line of therapy.
   2. Salvage chemoimmunotherapy followed by stem cell transplantation will be considered as 1 line of therapy.
   3. Any maintenance therapy will not be counted as a separate line of systemic therapy.
   4. Radiation with curative intent for localized DLBCL will not be counted as 1 line of therapy
6. Documented radiographic evidence of progressive DLBCL of the last line (or refractory DLBCL) prior to the first dosing.

Exclusion Criteria:

1. Female patients who are pregnant or lactating
2. DLBCL with mucosa-associated lymphoid tissue [MALT] lymphoma, or primary mediastinal (thymic) large B-cell lymphoma (PMBL)
3. Known central nervous system lymphoma or meningeal involvement (for dose expansion phase, patients with stable CNS disease could be considered).
4. Patients eligible for high-dose chemotherapy with autologous stem cell transplantation rescue (the Investigator must provide detailed documentation for ineligibility)
5. Use of any standard or experimental anti-DLBCL therapy (including radiation, chemotherapy, immunotherapy, radio-immunotherapy, or any other anticancer therapy) <21 days prior to Cycle 1 Day 1.
6. Autologous stem cell transplant (SCT) <6 months or prior allogeneic SCT, or CAR-T cell infusion <6 months prior to Cycle 1.
7. Major surgery within 4 weeks of the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
MTD | the last patient on study has completed 12 months of follow-up
  Maximum Tolerated Dose
RP2D | the last patient on study has completed 12 months of follow-up
  Recommended Phase 2 Dose

SECONDARY OUTCOMES:
ORR | the last patient on study has completed 12 months of follow-up
  Overall Response Rate
PFS | the last patient on study has completed 12 months of follow-up
  Progression Free Survival
DOR | the last patient on study has completed 12 months of follow-up
  Duration of Response
OS | the last patient on study has completed 12 months of follow-up
  Overall Survival
TTR | the last patient on study has completed 12 months of follow-up
  Time To Response
TTP | the last patient on study has completed 12 months of follow-up
  Time To Progression

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yu, Study Director — Medical Monitor
Locations (6):
- China (6):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The first Affiliated Hospital of China medical University, Shenyang, Liaoning